CLINICAL TRIAL: NCT02660866
Title: Excellence In Peripheral Artery Disease Thrombin Receptor Antagonist Intervention In Claudication Evaluation (XLPAD-TRACE Trial)
Acronym: XLPADTRACE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Subhash Banerjee, Chief, Cardiology Division, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: xlpadtrace
Record Dates: First submitted 2015-12-30; First posted 2016-01-21 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Peripheral Arterial Disease
Keywords: intermittent claudication; randomized controlled trial
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — vorapaxar

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMT+APT+Placebo (Placebo Comparator): Standard Medical Therapy (SMT): Presence of any two of the listed classes of agents [angiotensin converting enzyme inhibitor (ACEI), angiotensin receptor blocker (ARB), statin therapy and beta-blocker drugs] + ability to perform at least 15 min of home walking a day, at least 3 times/week, at ≥20 steps/min
  Background Antiplatelet Therapy (APT) :At least one aspirin dose within 5 days prior to randomization at 325 mg dose in aspirin naïve patients (0-5 days of prior aspirin use) or at least one aspirin dose within 5 days prior to randomization at 81 mg dose in patients on chronic (>5 days of prior use) aspirin therapy.
  Interventions: Drug: Placebo + background APT + SMT; Drug: Vorapaxar 2.08 mg/d + background APT + SMT.
- SMT+APT+Vorapaxar (Active Comparator): Standard Medical Therapy (SMT): Presence of any two of the listed classes of agents [angiotensin converting enzyme inhibitor (ACEI), angiotensin receptor blocker (ARB), statin therapy and beta-blocker drugs] + ability to perform at least 15 min of home walking a day, at least 3 times/week, at ≥20 steps/min
  Background Antiplatelet Therapy (APT) :At least one aspirin dose within 5 days prior to randomization at 325 mg dose in aspirin naïve patients (0-5 days of prior aspirin use) or at least one aspirin dose within 5 days prior to randomization at 81 mg dose in patients on chronic (>5 days of prior use) aspirin therapy.
  Vorapaxar: Vorapaxar 2.08mg/day
  Interventions: Drug: Placebo + background APT + SMT; Drug: Vorapaxar 2.08 mg/d + background APT + SMT.

INTERVENTIONS:
Drug: Placebo + background APT + SMT — Placebo drug therapy combined with standard medical therapy combined with Antiplatelet therapy (Aspirin therapy)
Drug: Vorapaxar 2.08 mg/d + background APT + SMT. — Vorapaxar 2.08 mg/d combined with standard medical therapy combined with Antiplatelet therapy (Aspirin therapy)

SUMMARY:
This is a Phase 4, randomized clinical trial to evaluate whether addition of Vorapaxar 2.08 mg daily vs. placebo daily on background antiplatelet therapy, prescribed for 6 months to patients with established peripheral artery disease (PAD) and Intermittent Claudication (IC) treated with standard medical therapy (SMT) would lead to an improvement in the peak walking time (PWT).

DETAILED DESCRIPTION:
Primary trial objective: To evaluate whether addition of Vorapaxar 2.08 mg daily vs. placebo daily on background antiplatelet therapy, prescribed for 6 months to patients with established PAD and IC treated with standard medical therapy (SMT) would lead to an improvement in the peak walking time (PWT)

Study endpoints Primary endpoint: Change from baseline to 6 months in the PWT on a graded treadmill test (GTT per Gardner protocol) between participants enrolled in the test and control arms of the study

Secondary endpoints

* Change from baseline to 6 months in the claudication onset time (COT) on GTT between participants enrolled in the test and control arms of the study.
* Change from baseline to 6 months in the walking impairment questionnaire distance scores (WIQ) between participants enrolled in the test and control arms of the study.
* Change from baseline to 6 months in self-reported quality of life score using the Medical Outcomes Study 12-Item Short form survey (SF-12) between participants enrolled in the test and control arms of the study

Tertiary endpoints

* The first occurrence of clinically indicated lower extremity endovascular or surgical revascularization procedure during the entire study duration post-randomization in participants enrolled in the test or control arms of the study.
* The first occurrence of all-cause death, MI, ischemic stroke during the entire study duration post-randomization in participants enrolled in the test or control arms of the study.
* The first occurrence of severe bleeding defined according to the Global Utilization of Streptokinase and Tissue plasminogen activator for Occluded coronary arteries (GUSTO) classification during the entire study duration post-randomization in participants enrolled in the test or control arms of the study.

ELIGIBILITY:
Pre-screening criteria

* Laboratory values available ≤ 1 year of the date of screening: hemoglobin ≥9g, platelet count >50,000 mm3 or <600,000 mm3
* No history of stroke or transient ischemic attack (TIA)
* No allergy to aspirin
* ≥40 years of age
* Presence of documented PAD by ABI <0.80 at rest or ≥20% drop in claudication limited exercise ABI in any limb and one of the following criteria in the corresponding limb:

  i.Prior surgical and/or endovascular lower extremity intervention (infra-renal aorta to pedal arteries) ii. Known presence of flow-limiting stenosis (≥70%) by clinically indicated angiography, computed tomographic (CT) or magnetic resonance imaging (MRI) tests or by Duplex ultrasonography (DUS) defined standard clinical criteria in lower extremity arteries
* Documented IC Rutherford/Becker (RC) category ≥2
* Presence of any one of the listed classes of agents [angiotensin converting enzyme inhibitor (ACEI), angiotensin receptor blocker (ARB), lipid lowering therapy, aspirin and beta-blocker drugs]-No MI or percutaneous coronary intervention (PCI) with DES within the past 11 months
* No planned surgical or endovascular procedures other than for the treatment of IC for the expected duration of the study
* No warfarin or other chronic oral anticoagulant use within the last 14 days
* No use of ticagrelor, clopidogrel, prasugrel or ticlopidine within last 7 days
* No contraindication(s) to the use of antithrombin or antiplatelet agents (history of intra-cerebral hemorrhage or ICH, presence of intracerebral mass, recent or <12 weeks gastrointestinal bleed requiring blood transfusion, any blood transfusion within the last 6 weeks, any trauma requiring surgery within the last 4 weeks or any surgical or endovascular procedure within the last 4 weeks
* No use of cilostazol and/or pentoxyphilline within last 7 days
* Severe psychiatric or behavioral illness that in the judgement of the investigator precludes study participation
* No history of major or minor amputation
* Severe heart, vascular and lung disease in the discretion of the investigator that precludes study participation.
* Ability to walk for at least 15 min/day, at least 3 days/week, at ≥20 steps/min

Inclusion criteria

* Treadmill PWT= 2-10 min on Gardner protocol
* Estimated survival ≥1 year in the judgment of the site investigator
* Use of at least one aspirin dose within at least 5 days prior to randomization at 325 mg dose in aspirin naïve patients (0-5 days of prior aspirin use) or at least one aspirin dose prior to randomization at 81 mg dose in patients on chronic (>5 days) aspirin therapy (at clinically indicated doses).
* Presence of any one of the listed classes of agents [angiotensin converting enzyme inhibitor (ACEI), angiotensin receptor blocker (ARB), lipid lowering therapy, aspirin and beta-blocker drugs]

Exclusion Criteria:

* MI or percutaneous coronary intervention (PCI) with DES within the past 11 months
* Positive pregnancy test
* Planned surgical or endovascular procedures other than for the treatment of IC
* Warfarin or other chronic oral anticoagulant use within 14 days
* Use of Ticagrelor, Clopidogrel, Prasugrel or Ticlopidine within 7 days
* Contraindication(s) to the use of antithrombin or antiplatelet agents (history of intra-cerebral hemorrhage or ICH, presence of intracerebral mass, recent or <12 weeks gastrointestinal bleed requiring blood transfusion, any blood transfusion within the last 6 weeks, any trauma requiring surgery within the last 4 weeks or any surgical or endovascular procedure within the last 4 weeks
* Use of cilostazol and/or pentoxyphilline within 7 days

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 6 months in the PWT on a graded treadmill test (GTT per Gardner protocol) between participants enrolled in the test and control arms of the study | 6 months

SECONDARY OUTCOMES:
Change from baseline to 6 months in the claudication onset time (COT) on GTT between participants enrolled in the test and control arms of the study. | 6 months
  Change from baseline to 6 months in the walking impairment questionnaire distance scores (WIQ) between participants enrolled in the test and control arms of the study.
  Change from baseline to 6 months in self-reported quality of life score using the Medical Outcomes Study 12-Item Short form survey (SF-12) between participants enrolled in the test and control arms of the study.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - San Diego VA Medical center, San Diego, California
  - VA Eastern Colorado Healthcare System, Denver, Colorado
  - Atlanta Heart Specialists, Atlanta, Georgia
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Minneapolis VA Medical center, Minneapolis, Minnesota
  - Creighton University, Omaha, Nebraska
  - Northwell Health, Manhasset, New York
  - OKlahoma VA Medical Center, Oklahoma City, Oklahoma
  - VA Portland Health Care System, Portland, Oregon
  - VA North Texas Health Care System, Dallas, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study results will be shared through clinicaltrials.gov and other publically available portals.

REFERENCES:
- [Result] Hirsch AT, Hiatt WR; PARTNERS Steering Committee. PAD awareness, risk, and treatment: new resources for survival--the USA PARTNERS program. Vasc Med. 2001;6(3 Suppl):9-12. doi: 10.1177/1358836X0100600i103. PMID 11789964
- [Result] McBurney CR, Eagle KA, Kline-Rogers EM, Cooper JV, Mani OC, Smith DE, Erickson SR. Health-related quality of life in patients 7 months after a myocardial infarction: factors affecting the Short Form-12. Pharmacotherapy. 2002 Dec;22(12):1616-22. doi: 10.1592/phco.22.17.1616.34121. PMID 12495171
- [Derived] Tsai S, Liu Y, Alaiti MA, Gutierrez JA, Brilakis ES, Banerjee S. No benefit of vorapaxar on walking performance in patients with intermittent claudication. Vasc Med. 2022 Feb;27(1):33-38. doi: 10.1177/1358863X211042082. Epub 2021 Oct 5. PMID 34609939